CLINICAL TRIAL: NCT06832709
Title: Etat Des Lieux De La Santé Physique, Sociale Et Psychologique Des Aidants Dans Le Cadre Des Maladies Respiratoires Chroniques
Brief Title: Fitness and Well-being of Caregivers in the Hauts-de-France Region
Acronym: PRHCARER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lille University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D2024-6
Record Dates: First submitted 2025-01-27; First posted 2025-02-18 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: caregivers; fitness; mental health; chronic respiratory disease
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Parallel assignment (2 groups)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- program of rehabilitation at home (Experimental): group of caregivers which their loved ones followed a program of rehabilitataion at home
  Interventions: Other: a program of rehabilitation
- a program of rehabilitation in a specialized center (Active Comparator): group of caregivers which their loved ones followed a program of rehabilitation in a specialized center
  Interventions: Other: a program of rehabilitation

INTERVENTIONS:
Other: a program of rehabilitation — physical activities, health education, psychosocial and motivational support

SUMMARY:
The ageing of the population is accompanied by an increase in the frequency of chronic illnesses, leading to a rise in the number of caregivers. These caregivers do not have the time to look after their own health, and they are very often in a deteriorated mental state with no knowledge of their level of fitness. A deterioration in their fitness can be a source of the development of diseases induced by a sedentary lifestyle. On the other hand, patients with chronic respiratory disease can benefit from respiratory rehabilitation (RR), which includes outpatient or home-based physical activity. The literature has demonstrated an improvement in the mental state of caregivers following a RR carried out by their loved ones without taking an interest in their fitness. The aim of the study will be to establish 1. a representation of the level of fitness and mental state of caregivers; 2. to assess the presence/absence of benefits on fitness and mental state of caregivers depending on the form of RR: home versus outpatient where the caregiver is not integrated in this last form.

DETAILED DESCRIPTION:
The literature reports more anxiety and depressive symptoms , a greater psychological and social burden and a poorer quality of life in caregivers than in their non-caregivers peers. Knowing the fitness of caregivers, by means of an assessment of their abilities, would make it possible to define their profile, which should reflect an altered fitness linked to a state of ill-being. The results of these assessments would make it possible to establish a prevention policy, and following a rehabilitation programme for their patients, their health should improve. For caregivers who agree to take part in the study, their physical, mental and social health will be assessed. The total duration of the visit, including all the assessments, is estimated at 1h30. We expect the fitness and mental and social state of all the caregivers to deteriorate in line with the indicators available in the literature for people of the same age who are not carers. Following care of the patients, we expect an improvement in fitness and mental state of the carers.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age;
* Have a sick relative taking part in a RR program, either as an outpatient at the Clinique de la Mitterie or at home with FormAction Santé;
* Have the cognitive ability to understand the instructions for carrying out the physical tests and the questions for answering the questionnaires;
* Be able to read;
* Have no disability preventing them from carrying out the physical tests;
* Have given their written consent to take part in the research;
* Be willing to comply with all the research procedures and duration.

Exclusion Criteria:

* Refusal to sign consent;
* Operation less than one month old;
* Presence of psychological or psychiatric disorders;
* Impossibility of receiving informed information;
* Impossibility of participating in the entire study;
* Contraindication to physical activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
functional capacity | 8 weeks
  achieve the highest number of steps on a stepper in 6 minutes

SECONDARY OUTCOMES:
assessments of fitness | 8 weeks
  handgrip
Short battery physical fitness test | 8 weeks
  SPPB (Short Physical Performance Battery) is the sum of the scores following 3 criteria: the balance test, the walking speed test and the chair rise test. This test makes it possible to evaluate an individual's physical performance.
  Score: 0 to 12 with best performance at 12.
Assessment of the state of health felt by the two parts of the EuroQol Group questionnaire (1990), | 8 weeks
  Test of: 5 questions offering a score between 1 and 5. Final score: 5 the best result, 15 the worst result.
  Helps to indicate how good or bad a state of health is, with a graduated scale (like that of a thermometer) on which 100 is the best state of health you can imagine and 0 is the worst state of health you can imagine. you can imagine.
  This scale is numbered from 0 to 100:
  * 100 is the healthiest imaginable.
  * 0 is the worst health imaginable.
Physical and mental fatigue questionnaire (Michielsen et al. 2003) | 8 weeks
  10 questions regarding the usual state. With 5 answer options ranging from "never (1)" to "always (5)" The total score is between 10 and 50. (10 = less fatigue, 50 = significant fatigue)
Charlson Comorbidity Score | 8 weeks
  Evaluates the level of comorbidity by considering the severity level of 19 predefined comorbidity disorders The investigator counts the number of points without indicating the items. Score 0 to 39 pts. 0 being the least and 39 being the serious
Visual analog scales to measure shortness of breath and fatigue felt in the legs | 8 weeks
  Two score scales ranging from 0 to 10 assessing the intensity of fatigue, shortness of breath and fatigue in the legs. 0 being the least serious and 10 being the highest fatigue.
Questionnaire on the Perceived Social Burden of Caregivers (Zarit et al., 1986) | 8 weeks
  22 questions on the different feelings of caregivers regarding their personal situations in the context of patient care.
  Answers ranging from never (0) to almost always (4) Total score ranging from 0 to 88 pts 0 being the most serious month and 88 being the most serious.
Anxiety and Depression Symptoms Questionnaire (Zigmond et al. 1983) | 8 weeks
  To detect anxious and depressive symptoms, the following interpretation can be proposed for each of the scores (A and D):
  Total score in 2 categories (A = anxiety and D = depression) 0 = least serious score 21 = worst score
EPICES social insecurity questionnaire (Sass et al. 2006) | 8 weeks
  questions on the means, assistance, leisure and housing of the caregiver. The score is continuous, it varies from 0 (absence of precariousness) to 100 (maximum of precariousness). The threshold of 30 is considered the precariousness threshold according to EPICES.

CONTACTS AND LOCATIONS:
Overall Officials: Claudine Fabre, PhD, Study Director — Lille University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Houben CHM, Spruit MA, Luyten H, Pennings HJ, van den Boogaart VEM, Creemers JPHM, Wesseling G, Wouters EFM, Janssen DJA. Cluster-randomised trial of a nurse-led advance care planning session in patients with COPD and their loved ones. Thorax. 2019 Apr;74(4):328-336. doi: 10.1136/thoraxjnl-2018-211943. Epub 2019 Jan 19. PMID 30661022
- [Background] Seamark DA, Blake SD, Seamark CJ, Halpin DM. Living with severe chronic obstructive pulmonary disease (COPD): perceptions of patients and their carers. An interpretative phenomenological analysis. Palliat Med. 2004 Oct;18(7):619-25. doi: 10.1191/0269216304pm928oa. PMID 15540670
- [Background] Grosbois JM, Gephine S, Kyheng M, Le Rouzic O, Chenivesse C. Improving the wellbeing of caregivers of patients with COPD using a home-based pulmonary rehabilitation programme. ERJ Open Res. 2022 Dec 12;8(4):00255-2022. doi: 10.1183/23120541.00255-2022. eCollection 2022 Oct. PMID 36655219